CLINICAL TRIAL: NCT04147598
Title: Dietary Control of Fat to Modify Colonic Inflammation in Ulcerative Colitis
Brief Title: Diet Study on Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Broad Medical Research Program Crohn's and Colitis Foundation (Unknown)
Responsible Party: Principal Investigator, Maria Abreu, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20130716
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory bowel disease; diet; low fat; UC; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Fat Diet (LFD) to Standard American Diet (SAD) (Experimental): Week 1 to 4 participants will receive a LFD followed by a washout period of 2 weeks and then week 6 to 10 SAD.
  Interventions: Other: LFD; Other: SAD
- SAD to LFD (Experimental): Week 1 to 4 participants will receive a SAD followed by a washout period of 2 weeks and then week 6 to 10 LFD.
  Interventions: Other: LFD; Other: SAD

INTERVENTIONS:
Other: LFD — Participants will receive daily prepared food trays to achieve a diet with approximately 10% of total fat, 1-5% of calories from saturated fat, and 5-9% of MUFA and PUFA. This diet will contain an approximate ratio of 1:1 of omega-6/omega-3 fatty acids.
Other: SAD — Participants will receive daily prepared food trays to achieve a diet with approximately 35-40% of calories from fat, 10-11% of saturated fats, and 25-29% would be mono-unsaturated (MUFA) and PUFA. This diet will contain a 20-30:1 ratio of omega-6/omega-3 fatty acids, representing the current SAD.

SUMMARY:
The primary purpose of this study is to determine the effectiveness of a low-fat or standard American diet (high in fat) in helping people with ulcerative colitis improve their symptoms and the signs of inflammation in blood tests and in bowel biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female ≥18 and ≤70 years old
2. History of UC of at least 3 months duration
3. UC should be confirmed by colonoscopy within two years of entry into the study
4. Patients with mild to moderate UC, or patients in remission that have had active disease within the past 18 months, regardless of treatment with mesalamines, immunosuppressants, anti-TNFs and/or vedolizumab

   * Patients on oral 5-aminosalicylates, mesalamine or sulfasalazine must be on a stable dose for ≥2 weeks prior to screening
   * Patients treated with anti-TNFs or immunosuppressants (AZA, 6-MP, or methotrexate) at screening must have been on a stable dose for ≥8 weeks and remain on the same dose during the treatment period
   * Patients on steroids can be on no more than prednisone 20mg daily or budesonide 9mg daily at screening. If clinically indicated, tapering of steroids after 4 weeks of intervention may occur. Prednisone may be tapered by no more than 2.5mg/week and budesonide by no more than 3mg/week.
   * Patients on infliximab, premedication may include intravenous corticosteroid
5. No antibiotic use or probiotic use within 4 weeks prior to screening
6. Signed written informed consent for enrollment into the study

Exclusion Criteria:

1. Patients with Crohn's Disease and Celiac Disease
2. History of colonic dysplasia except for adenoma on prior surveillance colonoscopy
3. Patients with altered anatomy: prior colectomy or anticipated colectomy during the study period and presence of ileal pouch or ostomy
4. Clinical manifestations concerning for fulminant disease or toxic megacolon
5. Patients with stool sample positive at during screening period or at least <12 weeks for ova, parasites, or culture for aerobic pathogens including: Aeromonas, Plesiomonas, Shigella, Yersinia, Campylobacter and E.coli spp. or positive for Clostridium difficile B toxin in stools
6. Use of cyclosporine, mycophenolate mofetil, sirolimus, thalidomide or tacrolimus within 2 months prior to screening
7. Need for prednisone >20mg daily or budesonide >9mg daily at the time of screening
8. Received intravenous corticosteroids within 2 weeks prior to screening, during screening, or during the study period, except as premedication for anti-TNFs
9. Use of Total Parenteral Nutrition at the time of screening and during the study period
10. Anti-diarrheal use within 2 weeks prior to screening
11. Presence of any of the following laboratory abnormalities during screening period or at least <12 weeks

    * Hemoglobin <8.0g/dl
    * Albumin <2.8g/dl
12. Conditions/situations such as:

    * Patients with short life expectancy
    * Uncooperative behavior or any condition that could make the patient potentially non-compliant to the study procedures
    * Patients with pacemaker
    * Other significant or life-threatening co-morbidities in which diet intervention could negatively affect
13. Failure to meet any of the inclusion criteria
14. Poor compliance with diet during the study period
15. Failure to submit stool samples as indicated at each phase of the study
16. The need for antibiotic use during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Change in quality of life as measured by the Short Inflammatory Bowel Disease Questionnaire (sIBDQ). | Baseline, 4 weeks
  sIBDQ is a 10-item shortened version of the original IBDQ assessing quality of life (QOL) with total scores ranging from 1 to 7 with a higher score indicating a better QOL.
Change in quality of life as measured by the Food-Related Quality of Life (FR-QoL-29) Questionnaire. | Baseline, 4 weeks
  FR-QoL-29 is a 29-item questionnaire assessing quality of life (QOL) with total scores ranging from 29 to 145 with a score less than 90 suggesting poor food related QoL.
Change in quality of life as measured by the Medical Outcomes Short Form-36 (SF-36) Questionnaire. | Baseline, 4 weeks
  SF-36 is a 36-item questionnaire assessing quality of life (QOL) with total scores ranging from 0 to 100 with a higher score indicating a better QOL.
Change in the expression of inflammatory markers in the colon. | Baseline, 4 weeks
  Change in the expression of interleukin (IL)-1β, IL-6 and Tumor Necrosis Factor alpha (TNFa) evaluated in pg/mL.
Change in the expression of cytokine in the colon. | Baseline, 4 weeks
  Change in the expression of cytokine high-sensitivity C-reactive protein (hsCRP) evaluted in mg/L.
Change in intestinal microbiota | Baseline, 4 weeks
  Change in relative abundance of the microbial communities evaluated as a percentage.

SECONDARY OUTCOMES:
Change in Ulcerative Colitis (UC) symptoms as measured by the partial Mayo score | Baseline, 4 weeks
  The partial Mayo score ranges from 0 to 9 with a higher score indicating worsening UC symptoms.
Change in UC symptoms as measured by the Simple Clinical Colitis Activity Index (SCCAI) | Baseline, 4 weeks
  SCCAI score ranges from 0 to 19 with a higher score indicating worsening UC symptoms.
Rate of adherence to fat intake | Baseline, 4 weeks
  Adherence to fat intake is measured by the web-based daily food diary software Nutrihand.
Rate of adherence to diet items | Baseline, 4 weeks
  Adherence to diet items is measured by the web-based daily food diary software Nutrihand.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Abreu, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fritsch J, Garces L, Quintero MA, Pignac-Kobinger J, Santander AM, Fernandez I, Ban YJ, Kwon D, Phillips MC, Knight K, Mao Q, Santaolalla R, Chen XS, Maruthamuthu M, Solis N, Damas OM, Kerman DH, Deshpande AR, Lewis JE, Chen C, Abreu MT. Low-Fat, High-Fiber Diet Reduces Markers of Inflammation and Dysbiosis and Improves Quality of Life in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1189-1199.e30. doi: 10.1016/j.cgh.2020.05.026. Epub 2020 May 20. PMID 32445952